CLINICAL TRIAL: NCT01314248
Title: A Randomized Crossover Comparison Between the Air-Q Intubating Laryngeal Airway the Laryngeal Mask Airway-Unique in Children
Brief Title: The Laryngeal Mask Airway (LMA) Unique and the Air-Q Intubating Laryngeal Airway (ILA) in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Attending, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: laryngeal mask airway & air Q
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Children
Keywords: airway sealing pressure; fiberoptic assessment; ease and time for successful insertion; incidence of gastric insufflation; complications were also evaluated

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- children weighing 10 to 15 kg
  Interventions: Device: each child will receive both the LMA and ILA

INTERVENTIONS:
Device: each child will receive both the LMA and ILA — each child will receive both the size 2 LMA and size 1.5 ILA

SUMMARY:
The air-Q® intubating laryngeal airway (ILA) is an supraglottic device used for both airway maintenance during routine anesthesia and as a conduit for tracheal intubation for patients with a difficult airway. The investigators goal for this study is to compare the performance of the ILA with the current standard of care the standard LMA during routine anesthesia.

DETAILED DESCRIPTION:
The goal for this randomized, crossover investigation is to compare a disposable version of the standard LMA, LMA Unique TM,with the air-Q ILA in pediatric patients. Oropharyngeal leak pressure is commonly used as an indicator of airway seal adequacy. Similarly, flexible fiberoptic bronchoscope examination is often employed to assess proper placement of airway devices. Our hypothesis is that the air-Q ILA is superior to the standard LMA in both these regards:

1. We hypothesize that airway leak pressures will be higher with the ILA. Airway leak pressures will be measured by recording the circuit pressure at which an equilibrium is reached.
2. We hypothesize that flexible fiberoptic view of the airway will be superior with the ILA. The airway view will be assessed using a previously used and published grading scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children undergoing general anesthesia using a supraglottic airway device
* 6 months to 36 months of age
* 10 to 15 kilograms in weight

Exclusion Criteria:

* Active respiratory infection
* History of difficult mask ventilation
* Features or history of a difficult airway
* Gastrointestinal reflux disease
* Clinically significant pulmonary disease

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children undergoing general anesthesia for their scheduled elective outpatient surgeries using a supraglottic airway device for airway maintenance.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Childrens Memorial Hospital
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Jagannathan N, Sohn LE, Mankoo R, Langen KE, Mandler T. A randomized crossover comparison between the Laryngeal Mask Airway-Unique and the air-Q intubating laryngeal airway in children. Paediatr Anaesth. 2012 Feb;22(2):161-7. doi: 10.1111/j.1460-9592.2011.03703.x. Epub 2011 Sep 15. PMID 21917058